CLINICAL TRIAL: NCT02737462
Title: A Phase I/II Study of CG200745 PPA to Determine the Maximum Tolerated Dose and Evaluate the Safety and Efficacy in Patients With Myelodysplastic Syndrome (MDS) Who Failed to Respond to Prior Hypomethylating Therapy
Brief Title: Phase 1/2 Study of CG200745 PPA for Myelodysplastic Syndrome
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: CrystalGenomics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CG200745-2-02
Record Dates: First submitted 2016-03-22; First posted 2016-04-14 (Estimated); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Myelodysplastic Syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — phosphoric acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CG200745 PPA (Experimental): CG200745 PPA intravenously daily for first 5 consecutive days per cycle (4 weeks)
  Interventions: Drug: CG200745 PPA

INTERVENTIONS:
Drug: CG200745 PPA — CG200745 PPA intravenously daily for first 5 consecutive days per cycle (4 weeks)
  Other Names: CG200745 PPA (phosphoric acid)

SUMMARY:
<Part I - Phase I trial> The phase I clinical trial is to identify the MTD (Maximum Tolerated Dose) and DLT (Dose Limiting Toxicity) of CG200745 PPA. Initial dose of CG200745 PPA is 150 mg/m^2, and it will be extended to 225 mg/m^2, 300 mg/m^2 or it will be reduced to 75 mg/m^2 based on the results of the cohort of 3 to 6 subjects per dose level.

Based on the 3+3 dose escalation study design, CG200745 PPA is to be administered according to the dose level. Each cohort consists of 3 or 6 subjects.

<Part II - Phase II trial> In the phase II clinical trial, the subjects will be administered with the dose which is to be identified as a recommended dose based on the results of Phase I study. Each cycle consisted of 28 days, same as the phase I. The entire treatment period is 6 cycles and tumor assessment is to be evaluated at the end of every 2 cycles.

DETAILED DESCRIPTION:
<Part I - Phase I trial> The phase I clinical trial is to identify the MTD and DLT of CG200745 PPA. Initial dose of CG200745 PPA is 150 mg/m^2, and it will be extended to 225 mg/m^2, 300 mg/m^2 or it will be reduced to 75 mg/m^2 based on the results of the cohort of 3 - 6 subjects per dose level.

Based on the 3+3 dose escalation study design, CG200745 PPA is to be administered as in four different cohorts according to the dose level. Each cohort consists of 3 or 6 subjects.

* Dose Level -1: CG200745 PPA 75 mg/m^2 x 5 (375 mg/m^2/cycle) / -50%
* Dose Level 1: CG200745 PPA 150 mg/m^2 x 5 (750 mg/m^2/cycle) / initial base dose
* Dose Level 2: CG200745 PPA 225 mg/m^2 x 5 (1,125 mg/m^2/cycle) / 50%
* Dose Level 3: CG200745 PPA 300 mg/m^2 x 5 (1,500 mg/m^2/cycle) / 33%

<Part II - Phase II trial> In the phase II clinical trial, the subjects will be administered with the dose which is to be identified as a recommended dose based on the results of Phase I study. Each cycle consisted of 28 days, same as the phase I. The entire treatment period is 6 cycles and tumor assessment is to be evaluated at the end of every 2 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Ages: 20 years and above
* Patient with MDS according to French-American-British (FAB) classification
* Patients who failed to respond to prior hypomethylating agents (5-azacytidine, decitabine)
* Eastern Cooperative Oncology Group (ECOG) performance status: 0-2
* Adequate renal and hepatic function

  * Total serum bilirubin ≤ 3 x Upper Limit Normal (ULN) (except for the case of increased unconjugated bilirubin)
  * Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), and Alkaline phosphatase (ALP) < 3 x ULN
  * Calculated Glomerular Filtration Rate (GFR) ≥ 50
* Fertile patients, except post-menopausal patients (no menstruation for at least 2 years) or proof of surgical sterility, must use effective contraception up to 3 months after the completion or withdrawal of the study.
* Negative pregnancy test
* Patients who understand the overall procedures and requirements of the study

Exclusion Criteria:

* Peripheral or bone marrow blasts: > 30%
* Less than 4 weeks since major surgery or radiotherapy
* Patient with clinically meaningful and relevant, active Central Nerve System (CNS) disorder
* Patient with active liver disease
* Patient with HIV positive
* Hyper-sensitivity to study drug or similar substances of the drugs
* Prior Histone Deacetylase (HDAC) inhibitor therapy
* Less than 4 weeks since hypomethylating agent or cytotoxic drug therapy
* Less than 4 weeks since immunosuppressive drug therapy
* Patient who participated in another clinical trial within past 4 weeks
* Patient who have severe diseases:

  * Severe cardiovascular diseases (severe or unstable angina, congestive heart failure, myocardial infarction within past 1 year, uncontrolled hypertension and uncontrolled arrhythmia)
  * Neurological or psychiatric disorder
  * Active uncontrolled infection
  * Any other diseases that may interfere with the interpretation of study result (according to the judgment of investigator)
* Pregnancy or lactating
* Patient who is not considered to be appropriate for the study according to the judgment of investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2016-06 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | up to 6 cycles (each cycle is 28 days)
  ORR is the proportion of the subjects with Complete Response (CR), Partial Response (PR), marrow CR (mCR), and hematological improvement (HI) in comparison to the total subjects

SECONDARY OUTCOMES:
Area Under the Curve [AUC] | Part I, Cycle 1, Day 1, up to 6 days
  Pharmacokinetics (PK) parameter
Maximum Plasma Concentration [Cmax] | Part I, Cycle 1, Day 1, up to 6 days
  Pharmacokinetics (PK) parameter
Adverse Event | up to 6 cycles
  Safety parameter
Clinical laboratory tests | up to 6 cycles
  Safety parameter

CONTACTS AND LOCATIONS:
Overall Officials: Je-Hwan Lee, M.D., PhD., Principal Investigator — Asan Medical Center; Jun Ho Jang, M,D., Ph.D., Principal Investigator — Samsung Medical Center; Sung-soo Yoon, M,D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Asan Medical Center, Samsung Medical Center, Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided